CLINICAL TRIAL: NCT04950309
Title: Characterization of an Optically Pumped Magnetometer (OPM) Magnetoencephalography (MEG) Array
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 210018; 21-M-0018
Record Dates: First submitted 2021-07-02; First posted 2021-07-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-25

CONDITIONS: Normal Physiology
Keywords: Imaging; biomagnetism; somatotopy; optically pumped magnetometer; Magnetoencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPM Array studies (Experimental): Testing of a final 49-61 channel OPM MEG system and any interim arrays
  Interventions: Device: SQUID MEG; Device: OPM MEG

INTERVENTIONS:
Device: SQUID MEG — MEG recordings acquired on a standard whole brain SQUID MEG system. Stimuli will be used, including auditory, visual, or somatosensory stimuli. Language stimuli and median nerve stimulation may also be used.
Device: OPM MEG — MEG recordings acquired on an investigational OPM MEG system. Stimuli will be used, including auditory, visual, or somatosensory stimuli. Language stimuli and median nerve stimulation may also be used.

SUMMARY:
Background:

Brain activity produces magnetic fields. These fields can be measured outside the head. Existing technology, called MEG, measures these fields. Researchers are testing a new type of magnetic field sensor called OPM. They hope it can help pinpoint with very high accuracy where brain activity is generated.

Objective:

To develop and test a new type of sensor for measuring the magnetic fields produced by brain activity.

Eligibility:

Healthy people ages 18-65 who had a magnetic resonance imaging (MRI) scan under protocol 17-M-0181.

Design:

Participants may be asked to complete sessions on both the traditional MEG instrument and the OPM array.

For the MEG, 3 small coils will be placed on the participant s face with tape. Their head will be positioned inside the MEG device.

For the OPM, sensors are housed in a 3d printed array. The sensors will be attached to a cap placed on the participant s head.

For both scans, participants will be seated in a chair inside a magnetically shielded room. They may complete several tasks. In one task, plastic cells will be placed on their fingers. Puffs of air will be sent to these cells, which will stimulate the sense of touch. Other tasks may include the following stimuli: visual (such as checkerboards), auditory (such as beeps and tones), or language (words and letters).

Researchers may also obtain recordings while they stimulate the nerve in the participant s forearm using electrical current in small electrodes.

Participation is expected to last for 1 day. Additional optional scans may be offered for up to 1 year....

DETAILED DESCRIPTION:
Study Description:

This protocol is a technical development protocol to characterize an optically pumped magnetometer (OPM) array used for measuring magnetic brain signals. We hypothesize that with our OPM arrays, we can achieve similar or better spatial resolution to that of a conventional MEG system.

Objectives:

Primary Objective 1: To fully characterize the performance of an OPM MEG array.

Primary Objective 2: To demonstrate that the OPM system can produce somatotopic maps accurately differentiating receptive fields of each finger. If successful, we will additionally determine if the system can differentiate receptive fields of each phalanx.

Endpoints:

Primary Endpoint: OPM array characterization parameters including signal to noise, sensitivity, bandwidth, and spatial

resolution, and comparison to similar parameters acquired on a standard SQID system.

Secondary Endpoint: Somatotopic representations of the digits of the hand

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-65
4. In good general health as evaluated according to protocol 17-M-0181
5. Completed a magnetic resonance imaging (MRI) scan under 17-M-0181

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Participants excluded from 17-M-0181 will be excluded from this protocol
2. Metal in the body which would cause artifacts on MEG recordings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
array characterization metrics | throughout protocol
  At each phase of array construction characterization parameters including signal to noise, sensitivity, bandwidth, and spatial resolution will be measured.

SECONDARY OUTCOMES:
Somatotopic representations | throughout protocol
  Somatotopic representations of the digits of the hand, potentially differentiating the individual phalanx of each finger.

CONTACTS AND LOCATIONS:
Overall Officials: Allison C Nugent, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
MEG datasets ultimately used for publication will be shared.
Supporting Information: Analytic Code
Time Frame: Data analysis code may be shared at the time of publication.
Access Criteria: Data will be shared without a specific DUA using an NIH supported online repository such as OpenNeuro.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-M-0018.html